CLINICAL TRIAL: NCT03491696
Title: Effects of the Addition of Metyrapone to Antidepressant Therapy in Depression With Dexamethasone Suppression Test Non-suppression.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Rouffach (Other)
Collaborators: University Hospital, Strasbourg, France (Other)
Responsible Party: Principal Investigator, Ludovic C. Jeanjean, Intern, Principal Investigator, Centre Hospitalier Rouffach
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A00628-47; 2018-000807-18 (EudraCT Number)
Record Dates: First submitted 2018-03-24; First posted 2018-04-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Depressive Disorder; Hormone Disturbance
Keywords: Depressive disorder; Metyrapone; Dexamethasone Suppression Test; Antidepressive association; Hypothalamic-pituitary-adrenal axis; Cortisol; Selective Serotonin Reuptake Inhibitor; Serotonin and Norepinephrine Reuptake Inhibitor
MeSH Terms: conditions — Depressive Disorder; Endocrine System Diseases | interventions — Metyrapone

STUDY DESIGN:
Intervention Model Description: It is an exploratory open label study with a single group, considered as a population of interest. Datas will be reported to existing knowledges and could not be a evidence of an effect but a suggestion for eventual future studies which have to be controlled versus placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): It is an open label study, designed with 14 patients, men and women, from 18 to 60 years old, hospitalized for a characterized depressive episode (as defined by International Classification of Diseases version 10 criteria). They have to be refractory to an antidepressant treatment prescribed in primary care medicine and have a Dexamethasone Suppression Test (DTS) non-suppression status. All patients included will take the association of SSRI/SNRI and METYRAPONE for 28 days.
  Interventions: Drug: Metyrapone

INTERVENTIONS:
Drug: Metyrapone — Association of Selective Serotonin Reuptake Inhibitor or Serotonin and Norepinephrine Reuptake Inhibitor and METYRAPONE. Duration of the association : 28 days.

SUMMARY:
The hypothesis of a link between depression and Hypothalamic-Pituitary Axis (HPA) dysfunction is now experienced. Since a first description in 1949 this link has made the HPA one of the most investigated hormonal axis in depression.

Many studies have demonstrated quantitative variations of circulating cortisol in situation of depression including increasing of basal concentration of blood cortisol or Adrenocorticotropic Hormone (ACTH). Furthermore there is an attenuated negative feedback performance of the blood cortisol on the release of ACTH and cortisol. This attenuation seems to be a consequence of a bluntness of sensibility of the hypothalamic cells and their Glucocorticoids Receptors type 2. Actually it seems that these phenomena are included in a diversion of the cortisol's action. From a function of acute stress management, with short-time exposures, the cortisol become one of the factors increasing an allostatic load, or resulting of this increase, maintaining a permanent state of stress, an inertia delay to adaptation and facilitating the emergence of psychiatric disorders.

This lack of function can be estimated by the Dexamethasone Suppression Test (DST) which, by stimulation attempting of feedback mechanisms by Dexamethasone (which has cortisol-like properties), can show a non-suppressor population with HPA bluntness. If this biological feature isn't a biological marker of depression, because of a lack of specificity and sensibility, is notably associated with a poor outcome and higher risks of suicidal behaviors and pharmacological resistance.

Many studies have explored possibilities of action on the HPA to treat depression or improve antidepressant specific therapeutics, with inconstant results. One of the most promising molecule seems to be Metyrapone, a reversible inhibitor of the 11ß-hydroxylase enzyme which transform desoxycorticosterone and 11deoxycortisol to respectively corticosterone and cortisol. There have been several open label studies which aim to explore the possibility of an effect of the combination between Metyrapone and antidepressant molecules. This led to two randomized double blind controlled versus placebo studies whose conclusions are divergent.

These conclusions and their heterogeneity lead to think that there is a sub-population which could be better responder to this type of association. Physiopathological knowledges and preliminary observations in DST non-suppressor population by using anti-glucocorticoids therapies , makes it possible to consider possible that responsive sub-population can be defined by the feature " DST non-suppressor ".

DETAILED DESCRIPTION:
Depression is now a public health issue, concerning 300 billion people in the World it is the leading cause of disability according to the World Health Organization and 800 000 persons die each year by committing suicide. Despite the finding of specific and efficiency treatments, recommended by main guidelines, a first prescription of antidepressant, Specific Serotonin Reuptake Inhibitor (SSRI) or Serotonin and Norepinephrine Reuptake Inhibitors (SNRI), is associated with a remission in only 35 to 45%. Using switch strategies in case of non-response and the fact that the number of antidepressant molecules stagnates from few decades lead patients to refractory disease and heavy care like using of mood-stabilizers molecules, Electro-Convulsive Therapy or Repetitive Trans-cranial Magnetic Stimulation. To avoid therapeutic escalation and limit collateral consequences it seems to be essential to understand physiopathological feature of each patient and proposing adapted treatment in front of early signs of resistance.

The hypothesis of a link between depression and Hypothalamic-Pituitary Axis (HPA) dysfunction is now experienced. Since a first description in 1949 this link has made the HPA one of the most investigated hormonal axis in depression.

Many studies have demonstrated quantitative variations of circulating cortisol in situation of depression including increasing of basal concentration of blood cortisol or Adrenocorticotropic Hormone (ACTH), a flattened rhythm of diurnal secretion, an early nadir and a disappearance of the morning secretion peak. Moreover it has be observed an anarchic rhythm and an increased amplitude of the secretion peaks. Furthermore there is an attenuated negative feedback performance of the blood cortisol on the release of ACTH and cortisol. This attenuation seems to be a consequence of a bluntness of sensibility of the hypothalamic cells and their Glucocorticoids Receptors type 2 (GR2). This bluntness seems to be consequence of genetic and epigenetic factors including maternal behaviors but also inflammation status with cytokines activation and abnormalities into the GR2 recycling process, with persistence of altered receptors.

Actually it seems that these phenomena are included in a diversion of the cortisol's action. From a function of acute stress management, with short-time exposures, the cortisol become one of the factors increasing an allostatic load, or resulting of this increase, maintaining a permanent state of stress, an inertia delay to adaptation and facilitating the emergence of psychiatric disorders.

This lack of function can be estimated by the Dexamethasone Suppression Test (DST) which, by stimulation attempting of feedback mechanisms by Dexamethasone (which has cortisol-like properties), can show a non-suppressor population with HPA bluntness. If this biological feature isn't a biological marker of depression, because of a lack of specificity and sensibility, is notably associated with a poor outcome and higher risks of suicidal behaviors and pharmacological resistance.

Many studies have explored possibilities of action on the HPA to treat depression or improve antidepressant specific therapeutics, with inconstant results. One of the most promising molecule seems to be Metyrapone, a reversible inhibitor of the 11ß-hydroxylase enzyme which transform desoxycorticosterone and 11deoxycortisol to respectively corticosterone and cortisol. There have been several open label studies which aim to explore the possibility of an effect of the combination between Metyrapone and antidepressant molecules. This led to two randomized double blind controlled versus placebo studies whose conclusions are divergent : if the study of Jahn et al. have showed a significative amelioration of clinical response, by association SSRI with Metyrapone, the Antiglucocorticoid Augmentation of Anti-Depressants in Depression (ADD) Study concluded that this improvement is not significative in clinical routine practice.

These conclusions and their heterogeneity lead to think that there is a sub-population which could be better responder to this type of association. Physiopathological knowledges and preliminary observations in DST non-suppressor population by using anti-glucocorticoids therapies, makes it possible to consider possible that responsive sub-population can be defined by the feature " DST non-suppressor ".

This is a multicenter, open-label study in 14 patients, men and women, aged 18 to 60 years, hospitalized following a characterized depressive episode, with alteration of the response by the hypothalamic-pituitary axis to the Dexamethasone restriction test and resistant to an antidepressant treatment proposed in primary care medicine. The main investigator centre will be the Rouffach Hospital Centre, the co-investigator centre will be the Strasbourg University Hospital (Hôpitaux Civils de Strasbourg).

Patients eligible for the study will present:

A characterized depressive episode defined according to International Classification of Diseases version 10 (ICD-10) criteria.

Persistent symptomatology despite treatment with a selective serotonin reuptake inhibitor or a well-conducted serotonin and norepinephrine reuptake inhibitor (inclusion score >18 on the Hamilton Depression Scale 17 items).

An alteration of the hypothalamic-pituitary response to the Dexamethasone Suppression Test (DST) defined by a non-suppression of cortisol production after taking 1mg of Dexamethasone (defined by a blood cortisol>120nmol/L at 8AM).

For the duration of the study, the psychotropic treatment previously prescribed (before admission) will remain unchanged.

This is an exploratory pilot study. The primary purpose is to assess the possibility of obtaining a normalized biological response to the Dexamethasone Suppression Test by the addition of short-term Metyrapone therapy to antidepressant therapy.

Secondary purposes are:

To determine if this effect is accompanied by a clinical improvement in depression defined by a sufficient decrease on the Hamilton Depression Scale 17 items (score below 18).

To determine if such an effect persists at distance (1 month) from taking Metyrapone without modifying the initial psychotropic treatment.

In the case of highlighting of a effect new study protocols, in particular controlled studies versus placebo, could be proposed.

The study will be conducted in a hospital setting and according to good clinical practice. It will include :

A pre-selection visit (at the beginning of hospitalisation) including a clinical examination (somatic and psychiatric), routine biological examinations, a review of medical and surgical history and previous and current treatments.

An evaluation of the hypothalamic-pituitary axis by a dynamic Dexamethasone Suppression Test, the interpretation of the results and their announcement to the patient by a physician.

An inclusion visit including verification of inclusion and exclusion criteria and a presentation of the study to the patient with consent (Day 0).

Treatment with Metyrapone 1 gram per day divided into four 250mg doses: in the morning at 8AM, at noon (12PM), in the evening at 6PM and at 10PM. This administration scheme was chosen because it has already been published in the literature in a similar context. Treatment will be given for 4 weeks without interruption and on a consistent dosing schedule (Day 2- Day 29).

Three evaluations of the hypothalamic-pituitary axis by a Dexamethasone Suppression Test (respectively at Day 17, Day 29 and Day 60), interpretation of the results and their announcement to the patient by a physician. The Day 29 evaluation is the only measure used for the primary outcome.

A final study visit including a psychiatric clinical examination. The decision to continue or modify psychotropic treatment will depend on the clinical situation observed.

ELIGIBILITY:
Inclusion Criteria:

* Present International Classification of Diseases version 10 (ICD-10) diagnostic criteria:

of moderate (F32.1) or severe depressive episode without psychotic symptoms (F32.2).

or recurrent depressive disorder, current moderate episode (F33.1) or current severe episode without psychotic symptoms (F33.2).

* Persistent symptomatology despite treatment with a selective serotonin reuptake inhibitor or a well-conducted serotonin and norepinephrine reuptake inhibitor (inclusion score >18 on the Hamilton-17 item scale (HAMDS-17)).
* Present an alteration of the hypothalamic-pituitary response to the Dexamethasone Suppression Test defined by a non-suppression of cortisol production (defined by a DST>120nmol/L at 8h).
* Have signed an informed consent to participate indicating a clear understanding of the study objectives and all procedures required by the study and agree to participate and abide by the requirements and restrictions inherent in the study.
* Have a body mass index between 18 and 25 kg/m2 included.
* Be affiliated to or beneficiary from a social security program.

Exclusion Criteria:

* Not being able to give free and informed consent (including patients with judiciary protection).
* Have a psychiatric condition other than characterized depression.
* For women: being pregnant as determined by a blood or urine pregnancy test or breastfeeding.
* Have an acute or chronic clinically significant disease that the investigator believes may interfere with patient safety during the study, or may place the patient at undue risk or interfere with the study objectives (particularly endocrinopathies, neuro-endocrinopathies or somatic conditions such as renal, adrenal or cardiac failure).
* Have a significant suicidal risk (RSD>5 scale).
* Previous treatment with carbamazepine, long-acting neuroleptics, monoamine oxidase inhibitors, electroconvulsive-therapy.
* Have recently taken (<15 days) any medication that occasionally interferes with neuroendocrine and hypothalamic-pituitary adrenal function: steroidal anti-inflammatory drugs, gluco/mineralo-corticoid analogues, potassium-saving diuretics, Mifepristone, Ketoconazole.
* Recent benzodiazepine consumption (defined as less than 5 times the half-life of the molecule concerned).
* Have a recent (<1 year) history of substance abuse or drug addiction.
* Drink more than 40 g/day (1 glass[25 cl] of beer with 3° alcohol=7.5 g ; or 1 glass[25 cl] of beer with 6° alcohol=15 g ; or 1 glass[12.5 cl] of wine with 10° alcohol=12 g ; or 1 glass[4cl] of aperitif with 42° alcohol=17 g).
* Have a recognized contraindication to Metyrapone including manifest adrenocortical insufficiency and hypersensitivity to Metyrapone or any of the excipients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-12-22 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Blood cortisol rate during a Dexamethasone Suppression Test after 28days of treatment by association METYRAPONE and antidepressant (Serotonin Selective Reuptake Inhibitor or Serotonin and Norepinephrine Reuptake Inhibitor). | day 29
  Test protocol is defined as proposed by Carroll et al. and as used in routine at the "Pôle 8-9" service at Rouffach's Hospital. It suppose :
  0h : Administration of 1mg of Dexamethasone orally. 8h - 16h - 23h : Blood Cortisol measure. The significative threshold of 120nmol/ml is defined, as used in previous studies of the research team.
  Included patients present a cortisol at 8AM > 120nmol/L, they are considered as "non-suppressor". Presenting a blood cortisol rate at 8AM <120nmol/L at day 29 is considered as a change to a "suppressor" status and is considered as better outcome.

SECONDARY OUTCOMES:
Changes from baseline in Hamilton Depression Scale 17 items with 28days of treatment by association METYRAPONE and antidepressant (Serotonin Selective Reuptake Inhibitor or Serotonin and Norepinephrine Reuptake Inhibitor). | day 0 (selection) ; day 17, day 29, day 60
  Clinical evaluation supervised by an investigator. 17 items, each score is summed to the total score. Total range : 0 to 54, higher value represent a severe disorder. Scores are classified as normal (<9), mild depression (10 to 13), mild to moderate depression (14 to 17), and moderate to severe depression (>17).
  In this study included patients with a baseline score >18, lower values is considered as better outcome.
Changes from baseline in Hamilton Anxiety Scale with 28days of treatment by association METYRAPONE and antidepressant (Serotonin Selective Reuptake Inhibitor or Serotonin and Norepinephrine Reuptake Inhibitor). | day 0 (selection) ; day 17, day 29, day 60
  Clinical evaluation supervised by an investigator. 14 Items. Each item is scored on a scale of 0 (not present) to 4 (severe) and summed to the total score, total score range of 0-56, higher value represent severe disorder, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Changes from baseline in Beck Depression Inventory with 28days of treatment by association METYRAPONE and antidepressant (Serotonin Selective Reuptake Inhibitor or Serotonin and Norepinephrine Reuptake Inhibitor). | day 0 (selection) ; day 17, day 29, day 60
  Clinical evaluation by the patient himself. 21 individual scale items are scored on a 4-point continuum (0=least, 3=most), summed to the totale score with a total score range of 0-63. Higher scores represent severe disorder.
Changes from baseline in Cortisol Blood Rates During a Dexamethasone Suppression Test with 28days of treatment by association METYRAPONE and antidepressant (Serotonin Selective Reuptake Inhibitor or Serotonin and Norepinephrine Reuptake Inhibitor). | day 0 (selection) ; day 17, day 29, day 60
  Test protocol is defined as proposed by Carroll et al. and as used in routine at the "Pôle 8-9" service at Rouffach's Hospital. It suppose :
  0h : Administration of 1mg of Dexamethasone orally. 8h - 16h - 23h : Blood Cortisol measure. The significative threshold of 120nmol/ml is defined, as used in previous studies of the research team.
  Included patients present a cortisol at 8AM > 120nmol/L, they are considered as "non-suppressor". Present a blood cortisol rate at 8AM <120nmol/L at day 29 is considered as a change to a "suppressor" status and is considered as a better outcome.
  The purpose of this monitoring is evaluate the kinetic of cortisol's control restitution and the stability of a phenomena.

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic C. Jeanjean, Intern, Principal Investigator — Centre Hospitalier de Rouffach
Locations (2):
- France (2):
  - Hopitaux Universitares de Strasbourg, Strasbourg, Bas Rhin
  - Centre Hospitalier de Rouffach, Rouffach, Haut Rhin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thase ME, Entsuah AR, Rudolph RL. Remission rates during treatment with venlafaxine or selective serotonin reuptake inhibitors. Br J Psychiatry. 2001 Mar;178:234-41. doi: 10.1192/bjp.178.3.234. PMID 11230034
- [Background] Cowen PJ. Not fade away: the HPA axis and depression. Psychol Med. 2010 Jan;40(1):1-4. doi: 10.1017/S0033291709005558. PMID 19335939
- [Background] Stetler C, Miller GE. Depression and hypothalamic-pituitary-adrenal activation: a quantitative summary of four decades of research. Psychosom Med. 2011 Feb-Mar;73(2):114-26. doi: 10.1097/PSY.0b013e31820ad12b. Epub 2011 Jan 21. PMID 21257974
- [Background] Linkowski P. Neuroendocrine profiles in mood disorders. Int J Neuropsychopharmacol. 2003 Jun;6(2):191-7. doi: 10.1017/S1461145703003407. PMID 12890312
- [Background] Pariante CM, Miller AH. Glucocorticoid receptors in major depression: relevance to pathophysiology and treatment. Biol Psychiatry. 2001 Mar 1;49(5):391-404. doi: 10.1016/s0006-3223(00)01088-x. PMID 11274650
- [Background] Gray JD, Kogan JF, Marrocco J, McEwen BS. Genomic and epigenomic mechanisms of glucocorticoids in the brain. Nat Rev Endocrinol. 2017 Nov;13(11):661-673. doi: 10.1038/nrendo.2017.97. Epub 2017 Sep 1. PMID 28862266
- [Background] Weaver IC, Cervoni N, Champagne FA, D'Alessio AC, Sharma S, Seckl JR, Dymov S, Szyf M, Meaney MJ. Epigenetic programming by maternal behavior. Nat Neurosci. 2004 Aug;7(8):847-54. doi: 10.1038/nn1276. Epub 2004 Jun 27. PMID 15220929
- [Background] Herbert J, Goodyer IM, Grossman AB, Hastings MH, de Kloet ER, Lightman SL, Lupien SJ, Roozendaal B, Seckl JR. Do corticosteroids damage the brain? J Neuroendocrinol. 2006 Jun;18(6):393-411. doi: 10.1111/j.1365-2826.2006.01429.x. PMID 16684130
- [Background] McEwen BS. Mood disorders and allostatic load. Biol Psychiatry. 2003 Aug 1;54(3):200-7. doi: 10.1016/s0006-3223(03)00177-x. PMID 12893096
- [Background] Carroll BJ, Feinberg M, Greden JF, Tarika J, Albala AA, Haskett RF, James NM, Kronfol Z, Lohr N, Steiner M, de Vigne JP, Young E. A specific laboratory test for the diagnosis of melancholia. Standardization, validation, and clinical utility. Arch Gen Psychiatry. 1981 Jan;38(1):15-22. doi: 10.1001/archpsyc.1981.01780260017001. PMID 7458567
- [Background] Ribeiro SC, Tandon R, Grunhaus L, Greden JF. The DST as a predictor of outcome in depression: a meta-analysis. Am J Psychiatry. 1993 Nov;150(11):1618-29. doi: 10.1176/ajp.150.11.1618. PMID 8214170
- [Background] Gallagher P, Malik N, Newham J, Young AH, Ferrier IN, Mackin P. Antiglucocorticoid treatments for mood disorders. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD005168. doi: 10.1002/14651858.CD005168.pub2. PMID 18254070
- [Background] Maric NP, Adzic M. Pharmacological modulation of HPA axis in depression - new avenues for potential therapeutic benefits. Psychiatr Danub. 2013 Sep;25(3):299-305. PMID 24048401
- [Background] Murphy BE, Ghadirian AM, Dhar V. Neuroendocrine responses to inhibitors of steroid biosynthesis in patients with major depression resistant to antidepressant therapy. Can J Psychiatry. 1998 Apr;43(3):279-86. doi: 10.1177/070674379804300307. PMID 9561317
- [Background] Rogoz Z, Skuza G, Wojcikowski J, Daniel WA, Wrobel A, Dudek D, Zieba A. Effect of metyrapone supplementation on imipramine therapy in patients with treatment-resistant unipolar depression. Pol J Pharmacol. 2004 Nov-Dec;56(6):849-55. PMID 15662100
- [Background] Jahn H, Schick M, Kiefer F, Kellner M, Yassouridis A, Wiedemann K. Metyrapone as additive treatment in major depression: a double-blind and placebo-controlled trial. Arch Gen Psychiatry. 2004 Dec;61(12):1235-44. doi: 10.1001/archpsyc.61.12.1235. PMID 15583115
- [Background] McAllister-Williams RH, Anderson IM, Finkelmeyer A, Gallagher P, Grunze HC, Haddad PM, Hughes T, Lloyd AJ, Mamasoula C, McColl E, Pearce S, Siddiqi N, Sinha BN, Steen N, Wainwright J, Winter FH, Ferrier IN, Watson S; ADD Study Team. Antidepressant augmentation with metyrapone for treatment-resistant depression (the ADD study): a double-blind, randomised, placebo-controlled trial. Lancet Psychiatry. 2016 Feb;3(2):117-27. doi: 10.1016/S2215-0366(15)00436-8. Epub 2015 Dec 23. PMID 26727041
- [Background] Duval F, Mokrani MC, Erb A, Gonzalez Opera F, Calleja C, Paris V. Relationship between chronobiological thyrotropin and prolactin responses to protirelin (TRH) and suicidal behavior in depressed patients. Psychoneuroendocrinology. 2017 Nov;85:100-109. doi: 10.1016/j.psyneuen.2017.07.488. Epub 2017 Jul 28. PMID 28843902